CLINICAL TRIAL: NCT04613856
Title: Water Bolus Volumes During Continuous Exercise in Heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003387
Record Dates: First submitted 2020-10-30; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Dehydration (Physiology); Hyperthermia
MeSH Terms: conditions — Dehydration; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Randomized, counterbalanced, crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current Best Practice - 237 mL water bolus (Active Comparator)
  Interventions: Other: Hydration protocol - 237 mL water bolus
- New Intervention - 500 mL water bolus (Experimental)
  Interventions: Other: Hydration protocol - 500 mL water bolus

INTERVENTIONS:
Other: Hydration protocol - 237 mL water bolus — Subjects consume 237 mL of water every 20 minutes during 2 hours of high intensity work in the heat.
  Arms: Current Best Practice - 237 mL water bolus
Other: Hydration protocol - 500 mL water bolus — Subjects consume 500 mL of water every 40 minutes during 2 hours of high intensity work in the heat.
  Arms: New Intervention - 500 mL water bolus

SUMMARY:
Hydration is important to all individuals including occupational workers who complete physical activity in the heat. Current best practice guidelines suggest drinking a cup of water every 15-20 minutes during activity in a hot environment, but research shows this may not be ideal for best maintaining hydration. The goal of this study is to determine if larger, more frequent water boluses better maintain hydration than smaller, less frequent water boluses during moderate intensity physical activity in the heat.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-39 y old
* Self-reported to be healthy

Exclusion Criteria:

* Female
* Not within defined age range
* History of any cardiovascular, neurologic, or metabolic disease
* Current tobacco use or regular use within the last 2 years.
* Taking medications with known thermoregulatory or cardiovascular effects (e.g., aspirin, beta blockers, diuretics, psychotropics, etc.)
* Inability to follow the rules of the protocols or understand the consent form

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Percent body mass loss | 2 hours
  Percent body mass loss after water intake
Core temperature | 2 hours
  Core temperature after water intake

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research and Exercise in Special Environments, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD data can be provided upon written request.